CLINICAL TRIAL: NCT04323943
Title: Comparison of Thermo-plastic Versus Carbon Foot Ankle Orthosis to Improve Gait and Reduce Fatigue in Post-stroke Patients: a Biomechanical and Neurophysiological Study
Acronym: MECASPRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Collaborators: University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC28; ANSM (Other: 2019-A02957-50)
Record Dates: First submitted 2020-03-19; First posted 2020-03-27 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Hemiparesis;Poststroke/CVA; Gait, Hemiplegic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, open labelled, monocentric, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbon-AFO (C-AFO) (Experimental): Manufactured carbon ankle foot orthosis (C-AFO) Sprystep (Thuasne) will be provided to patients. A familiarization with C-AFO will be performed before doing the tests.
  Interventions: Device: Ankle Foot orthosis (AFO)
- Custom-made thermo-plastic orthosis (CM-AFO) (Active Comparator): Own custom-made thermo-plastic orthosis (CM-AFO) of patients. A familiarization will be performed also before doing the tests.
  Interventions: Device: Ankle Foot orthosis (AFO)
- Without orthosis (NO) (No Intervention): No orthosis - patient will wear only their shoes

INTERVENTIONS:
Device: Ankle Foot orthosis (AFO) — The experimental protocol will require 4 visits: one inclusion visit and 3 visits for evaluations. Each visit corresponds to one condition: C-AFO, CM-AFO or NO (according to a random order).
  Visit #1 will consist in a clinical evaluation and a familiarization session with the measuring devices and methodologies used in visit#2 #3 and #4.
  During #2, #3 and #4 visits (14 days between each session), the subject will perform with C-AFO, CM-AFO or NO according to the random order :
  * 5 x 15m overground at a comfortable walking speed (CWS) where EMG, ground reaction force and kinematics will be measured
  * 6MWT where energy cost will be measured
  * 5 x 15m overground (immediately after the 6MWT) at a comfortable walking speed
  Other Names: Sprystep (Thuasne)
  Arms: Carbon-AFO (C-AFO); Custom-made thermo-plastic orthosis (CM-AFO)

SUMMARY:
Approximately 20% of stroke survivors have difficulties to dorsiflex the ankle and clear the ground during walking. This impairment, termed as "foot drop", is caused by an association of weak dorsiflexors and increased spasticity and stiffness of the plantar-flexors. As a consequence, walking performances are reduced and energy cost of walking is deteriorated. This may increase performance fatigability, as the locomotion will be realized at a higher percentage of the subjects' capacities. In order to overcome these issues, different treatments are proposed. One of the most conventional solutions are the use of ankle foot orthosis (AFO) and it is the most commonly prescribed device used to compensate for "foot drop". There is a very large choice of AFO on the market which can be proposed to patients with foot drop.

The aim of this study is thus to assess the mechanical effects of using a manufactured carbon AFO in by comparison to a custom-made thermo-plastic AFO on walking capacity (distance and energy cost), fatigue and "foot drop" control throughout the gait phase in patients with hemiparetic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic patients, walking with CM-AFO
* Diagnosis of a first stroke since at least 6 months with medical conditions of stroke known, treatment proposed, cardio-vascular and neurological state stabilized
* Foot drop observed during the swing phase of gait, requiring the use of a custom-made plastic orthosis that has been used for at least 3 months and used for less than 2 years
* Muscle spasticity not higher than grade 3 according to the Modified Ashworth Scale
* Sufficient motor ability and endurance to ambulate at least 15 m independently without AFO
* Patient who signed a consent
* Patients affiliated or entitled to a social security system.

Exclusion Criteria:

* Patients who did not have brain MRI imaging after their stroke to confirm the diagnosis of stroke,
* Patients with an associated cerebellar syndrome,
* Patients with clinical brainstem involvement (cranial pair deficit),
* Patients with a neurological history other than stroke that has an impact on walking,
* Patients with unstable cardiovascular or respiratory disorders likely to induce gait disorders that may influence the performance of the tests to a greater extent than in the case of vascular hemiplegics,
* Patients with alcohol or drug dependence,
* Patients with psychiatric illness, cognitive impairment, uncontrolled disease/epilepsy, malignant pathology, renal impairment, unstable or decompensated diabetes, severe,
* Patients with a history of associated disabling systemic disease,
* Patients who refused to sign the written consent,
* Patients with a current pregnancy,
* Patients under court protection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Distance walked during the 6 Minute Walk Test (6MWT) | Day : 14
  Patient will performed three experimental session (14 days between each session) during wich the primary outcome will be assessed : one session while walking with C-AFO, one session while walking with CM-AFO, and one session while walking without AFO (randomized order).
  6 Minute Walk Test is a beneficial tool to evaluate walking endurance in patients with poststroke hemiparesis

SECONDARY OUTCOMES:
Energy cost | Day : 14
  Energy cost will be assessed by oxygen consumption recorded during the 6MWT in the 3 conditions (C-AFO, CM-AFO, NO)
Muscular activity | Day: 14
  Muscular activity will be assessed by electromyography (EMG) on different muscles (anterior tibial, gastroc medial, femoral). Muscular activity will be assessed before and after 6MWT during 5*15m sessions
Angle | Day : 14
  Angle (°) of ankle, knee and hip will be assessed in the 3 conditions before and after 6MWT during 5*15 m sessions
Perceived fatigue | Day : 14
  Perceived fatigue will be assessed by the Rated Perceived Exertion (RPE) scale before and after 6MWT. The RPE scale runs from 0 - 10. 0 is related to an easy activity and 10 (very, very heavy) is related to a very difficult activity.
Power | Day : 14
  Power (watt) of ankle, knee and hip will be assessed in the 3 conditions before and after 6MWT during 5*15 m sessions
Momentum | Day : 14
  Momemtum (J rad-1) of ankle, knee and hip will be assessed in the 3 conditions before and after 6MWT during 5*15 m sessions
Satisfaction related to the device | Day : 42
  A satisfaction survey will be asked in order to assess the positioning of AFO, comfort, esthetic and global satisfaction of devices

CONTACTS AND LOCATIONS:
Overall Officials: Paul Calmels, MD,PhD, Principal Investigator — CHU Saint Etienne, Bellevue
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France